CLINICAL TRIAL: NCT00944359
Title: Community-based Intervention Trial to Compare the Impact of Preventive and Therapeutic Zinc Supplementation Programs Among Young Children in Burkina Faso
Brief Title: Impact of Preventive and Therapeutic Zinc Supplementation Programs Among Young Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Université Polytechnique de Bobo-Dioulasso (Other); Helen Keller International (Other); Thrasher Research Fund (Other); Canadian International Development Agency (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 222218; Zinc 7-20
Record Dates: First submitted 2009-07-21; First posted 2009-07-23 (Estimated); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: Zinc Deficiency; Diarrhea; Malaria
Keywords: zinc supplementation; diarrhea management; zinc deficiency; malaria
MeSH Terms: conditions — Diarrhea; Malaria

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Daily preventive Zn; placebo treatment (Experimental): 7 mg zinc per day for 12 months and placebo supplement during diarrhea episode
  Interventions: Dietary Supplement: Daily preventive Zn; placebo treatment
- Therapeutic Zn; daily placebo (Experimental): 20 mg of zinc for 10 days during episodes of diarrhea and daily placebo supplement
  Interventions: Dietary Supplement: Therapeutic Zn; daily placebo
- Intermittent Zn; placebo treatment (Experimental): 10 mg zinc for 10 days every 3 months, daily placebo during 80 days of 3 months period and placebo during diarrhea episode
  Interventions: Dietary Supplement: Intermittent Zn; placebo treatment
- Surveillance control group (Active Comparator): Surveillance control group will be randomly assigned to intervention groups every 3 months
  Interventions: Other: Surveillance control group
- Non-intervention (No Intervention): Standard care provided by health system

INTERVENTIONS:
Dietary Supplement: Daily preventive Zn; placebo treatment — 7 mg zinc / day and placebo supplement during diarrhea episodes
  Other Names: Nutriset preventive zinc and therapeutic placebo supplement
  Arms: Daily preventive Zn; placebo treatment
Dietary Supplement: Therapeutic Zn; daily placebo — 20 mg zinc / day for 10 days during diarrhea episodes and daily placebo supplement
  Other Names: Nutriset ZinCfant
  Arms: Therapeutic Zn; daily placebo
Dietary Supplement: Intermittent Zn; placebo treatment — 10 mg zinc for 10 days every 3 months, placebo supplements daily for all other days during 12 months; placebo supplements during diarrhea episodes
  Other Names: Nutriset zinc supplement
  Arms: Intermittent Zn; placebo treatment
Other: Surveillance control group — Active weekly morbidity surveillance for 3 months. New surveillance control group will be randomly assigned to intervention groups every 3 months
  Arms: Surveillance control group

SUMMARY:
Zinc supplementation can either be provided in a lower daily dose to prevent zinc deficiency or in a higher dose for 10-14 days as part of the treatment of diarrhea. It is important to determine how best to integrate programs designed either to prevent zinc deficiency or to treat diarrhea.

The overall objective of this project is to determine the most effective approach to prevent zinc deficiency and treat diarrhea, such that a single approach could provide the maximal beneficial impact on the health and nutritional status of young children and greatest simplicity of implementation.

DETAILED DESCRIPTION:
This is a single-center cluster- and household-randomized, partially masked, community-based efficacy trial of zinc supplementation. The study sample consists of 5 study groups in one region, with 34 clusters randomly assigned to 3 types of intervention communities.

Communities will be randomly assigned to 1) early intervention communities, 2) later intervention communities, 3) non-intervention communities. Within each intervention cluster, children will be randomly assigned to the intervention group at the household level. Children aged 6-27 months at enrollment will be eligible. The study duration is 12 months.

The investigators will assess the relative impact of daily preventive zinc supplementation (7 mg zinc/d for one year), intermittent preventive supplementation (10 mg zinc/d for 10 days every three months for one year), and zinc treatment during episodes of diarrhea (20 mg zinc/d for 10 days beginning with each episode of diarrhea during one year). Outcomes that will be assessed include the incidence and duration of all episodes of diarrhea, the incidence of malaria, physical growth, and (in a sub-group) biochemical indicators of zinc, iron and vitamin A status.

ELIGIBILITY:
Inclusion Criteria:

* 6-27 months of age
* Plan to remain in study area for 1 year

Exclusion Criteria:

* Evidence of congenital abnormalities and chronic infection
* Severe anemia and severe acute malnutrition
* Consumption of micronutrient supplementation including zinc

Ages: 6 Months to 27 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 7680 (Actual)
Dates: Start 2010-12; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Change in length and length-for-age Z-score | 12 months
Change in weight and weight-for-age | 12 months
Incidence of diarrhea and laboratory-confirmed malaria | 12 months
Change in plasma zinc concentration | 12 months

SECONDARY OUTCOMES:
Incidence of stunting, underweight, and wasting | 12 months
Change in hemoglobin and iron status | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth H Brown, MD, Principal Investigator — University of California, Davis
Locations (1):
- Institut de Recherche en Science de la Sante, Bobo-Dioulasso, Burkina Faso

REFERENCES:
- [Result] Becquey E, Ouedraogo CT, Hess SY, Rouamba N, Prince L, Ouedraogo JB, Vosti SA, Brown KH. Comparison of Preventive and Therapeutic Zinc Supplementation in Young Children in Burkina Faso: A Cluster-Randomized, Community-Based Trial. J Nutr. 2016 Oct;146(10):2058-2066. doi: 10.3945/jn.116.230128. Epub 2016 Aug 3. PMID 27489011
- [Result] Hess SY, Peerson JM, Becquey E, Abbeddou S, Ouedraogo CT, Some JW, Yakes Jimenez E, Ouedraogo JB, Vosti SA, Rouamba N, Brown KH. Differing growth responses to nutritional supplements in neighboring health districts of Burkina Faso are likely due to benefits of small-quantity lipid-based nutrient supplements (LNS). PLoS One. 2017 Aug 3;12(8):e0181770. doi: 10.1371/journal.pone.0181770. eCollection 2017. PMID 28771493
- [Derived] Imdad A, Rogner J, Sherwani RN, Sidhu J, Regan A, Haykal MR, Tsistinas O, Smith A, Chan XHS, Mayo-Wilson E, Bhutta ZA. Zinc supplementation for preventing mortality, morbidity, and growth failure in children aged 6 months to 12 years. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD009384. doi: 10.1002/14651858.CD009384.pub3. PMID 36994923